CLINICAL TRIAL: NCT04030741
Title: Non Operative Treatment With Antibiotics Vs Surgery for Acute Non Perforated Appendicitis in Children: A Randomized Controlled Trial.
Brief Title: Non-operative Treatment of Acute Non-perforated Appendicitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Fatima Numeri, Assistant Professor, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201/RC/KEMU
Record Dates: First submitted 2019-03-01; First posted 2019-07-24 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Acute Appendicitis
Keywords: Acute Appendicitis.; Pediatric Appendicitis Score (PAS).; Visual Analogue Scale (VAS) Score.
MeSH Terms: conditions — Appendicitis | interventions — Meropenem; Metronidazole; Appendectomy

STUDY DESIGN:
Intervention Model Description: After permission from the ethical review board (ERB), Children diagnosed with acute appendicitis and fulfilling the inclusion and exclusion criteria will be included in the study after taking informed consent from parents. All the patients inducted in the study will be randomly divided into two groups: Non-operative treatment (group A) and operative treatment (group B), using computer generated number. Total sample size is 180 patiens and duration is 3 to 6 months.
Masking Description: The individual who evaluates the outcome(s) of interest
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Meronem and flagyl (Active Comparator): Children in Non-operative treatment (group A) Children in non-operative treatment group will be given intravenous meropenem (10 mg/kg/dose x IV x TDS) and metronidazole (20 mg/kg/day divided into 3 doses) for at least 48 hours. Once the child starts tolerating oral intake and becomes clinically improved, the treatment will be changed to oral ciprofloxacin (20 mg/kg/day) divided into 2 divided doses) and metronidazole (20 mg/kg/day divided into 3 doses for another 8 days.
  Interventions: Drug: Meronem and flagyl
- Surgery (appendectomy) (Active Comparator): Children in group B: appendectomy will b done and post operative single dose of antibiotics.
  discharge after 24hour and Follow up after 1 week.
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Drug: Meronem and flagyl — meronem and flagy
  Other Names: Flagyl
  Arms: Meronem and flagyl
Procedure: Appendectomy — Appendectomy as treatment for acute appendicitis
  Arms: Surgery (appendectomy)

SUMMARY:
Gold Standard treatment of appendicitis is appendectomy but non-operative treatment of non-perforated appendicitis with antibiotics is also under trial. Although appendectomy is curative but it is an invasive procedure done under general anesthesia with different risks and complications during and after operation, leading to disturbance of child daily routines and activities. Reported rates of perioperative complications are from 5% - 10%, with serious complications occurring in 1% to 7% of patients.

Children presenting with acute (<2 days) right iliac fossa pain with pediatric appendicitis score >7, with none of the following on ultrasonography: abscess formation, or loss of the echogenic sub-mucosal layer of the appendix or presence of an appendicolith or periappendiceal fluid collection will be labeled as having appendicitis.

After diagnosis we divided the patients into two groups.patients in group A will be treated with antibiotics and appendectomy is done for group B patients.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common presenting conditions in pediatric emergencies. It has an estimated lifetime risk of about 8%. Although it commonly occurs in the second decade of life but 11.4% children are diagnosed with acute appendicitis in the pediatric emergency.

The rationale of my study is that limited local clinical trial is available regarding the efficacy of non-operative treatment with antibiotics vs operative treatment of acute non-perforated appendicitis in children.

All children between 5 and 15 years of age of both genders admitted in the pediatric surgery emergency with having pediatric appendicitis score (PAS anexure 1) >7 will be included in the study.

All the patients inducted in the study will be randomly divided into two groups: Non-operative treatment (group A) and operative treatment (group B), using computer generated number. Each patient will be evaluated and relevant data according to the predesigned questionnaire will be collected and documented. Age, duration of symptoms, body temperature,C-reactive protein, white blood cell, neutrophil concentrations, Ultrasound findings and PAS score will be noted at the time of admission. Children in non-operative treatment group will be given intravenous meropenem (10 mg/kg/dose x IV x TDS) and metronidazole (20 mg/kg/day divided into 3 doses) for at least 48 hours. Once the child starts tolerating oral intake and becomes clinically improved, the treatment will be changed to oral ciprofloxacin (20 mg/kg/day divided into 2 divided doses) and metronidazole (20 mg/kg × 1 per 24 hours) for another 8 days. Supportive care will be given equally to all the patients as protocol of treatment with regular vital monitoring. Improvement or development of complications will be noted. Discharge criteria for both groups will be: afebrile for 24 hours, with or without oral antibiotics, adequate pain relief on oral analgesia assesd by visual analogue scale ( VAS) scale (anexure 2), tolerating a light diet, and mobile.

Failure of non-operative treatment will be defined if any one of the following is seen: abscess formation or complex peri-appendiceal fluid collection seen on ultrasonography, the need for surgery (due to worsening of symptoms evaulated by history, physical examination and repeat ultrasonography) within 48 hours, or recurrence of appendicitis within 3 months.

Patients with recurrence of symptoms of appendicitis (right iliac fossa pain with pediatric appendicitis score >7) after complete resolution previously with non-operated treatment, will be labeled as Recurrent appendicitis.All the data will be collected on a preformed questionnaire. Discharge criteria for both the groups will be: afebrile for 24 hours, with or without oral antibiotics, adequate pain relief on oral analgesia and tolerating a light diet. Patient will be kept on follow-up in group-A for duration of 3 month to 6 month. Patients will be kept on follow-up in Outdoor patients department once in a week till 3 months in group B.

ANNEXURE 1: Pediatric Appendicitis Score (PAS)

No Symptoms Score

1. Right iliac fossa tenderness to cough, percussion, or hopping 2
2. Migration of pain to Right iliac fossa 1
3. Anorexia 1
4. Fever (Temperature ≥38.0ºC/100.4ºF) 1
5. Nausea or vomiting 1
6. Tenderness over right iliac fossa 2
7. Leukocytosis (WBC >10,000 ) 1
8. Left shift (PMN >7,500 ) 1

Acute Appendicitis if score is >7

Anexure 2 Visual Analogue Scale

0 = Relaxed and comfortable 1-3 = Mild discomfort 4-6 =Moderate pain 7-10 =Severe discomfort or pain or both

ELIGIBILITY:
Inclusion Criteria:

• All children between 5 and 15 years of age of both genders admitted in the pediatric surgery emergency with having PAS score >7will be included in the study.

Exclusion Criteria:

* Patient with suspicion of perforated appendicitis on the basis of generalized peritonitis and abscess formation on ultrasound.
* Patients with an appendicular mass, diagnosed by clinical examination and ultrasonography.
* Patient with previous non-operative treatment of acute appendicitis (recurrent appendicitis)
* Patients with C-reactive proteins > 40 mg/L.
* Patients with history of any previous abdominal surgery.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pain relief | 24 hour
  Pain relief assessed by visual analogue scale (VAS) score < 3
Afebrile | 24 hours
  Temperature less than 98 Fahrenheit.
Food Tolerance | 24 hour
  Child starts oral intake and had no symptoms after food intake.

SECONDARY OUTCOMES:
Recurrence of symptoms of acute appendicitis | Within 3 months.
  Child presented pain in right iliac fossa, nausea and loss appetite with PAS Score greater than 7.
  on examination: Tenderness and Rebound tenderness

CONTACTS AND LOCATIONS:
Overall Officials: Paediatric surgery department, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
First i have to publication of article then i want to make available for others.

REFERENCES:
- [Result] Di Saverio S, Birindelli A, Kelly MD, Catena F, Weber DG, Sartelli M, Sugrue M, De Moya M, Gomes CA, Bhangu A, Agresta F, Moore EE, Soreide K, Griffiths E, De Castro S, Kashuk J, Kluger Y, Leppaniemi A, Ansaloni L, Andersson M, Coccolini F, Coimbra R, Gurusamy KS, Campanile FC, Biffl W, Chiara O, Moore F, Peitzman AB, Fraga GP, Costa D, Maier RV, Rizoli S, Balogh ZJ, Bendinelli C, Cirocchi R, Tonini V, Piccinini A, Tugnoli G, Jovine E, Persiani R, Biondi A, Scalea T, Stahel P, Ivatury R, Velmahos G, Andersson R. WSES Jerusalem guidelines for diagnosis and treatment of acute appendicitis. World J Emerg Surg. 2016 Jul 18;11:34. doi: 10.1186/s13017-016-0090-5. eCollection 2016. PMID 27437029
- See also: Maggiore Hospital, AUSL, Bologna, Italy — https://www.ncbi.nlm.nih.gov/pubmed/27437029